CLINICAL TRIAL: NCT03772301
Title: Evaluation of Hoarding Behaviour and Eating Disorders Among Holocaust Survivors and Their Descendants
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: HYMC-0083-18
Record Dates: First submitted 2018-12-10; First posted 2018-12-11 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Hoarding Disorder
MeSH Terms: conditions — Hoarding Disorder

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: At least 200 Jewish Holocaust survivors of the first generation living in Germany and Israel - an equal number in each country
- Group 2: The second generation, whose parents lived in Europe during the Second World War, now live in Germany (originating from Western and Eastern Europe) - at least 200 participants.
- Group 3: Third generation of Jewish Holocaust survivors who participated in the first phase, currently living in Germany and Israel - at least 200 participants including at least 100 subjects in each country. These are adults only. The research program does not include children and adolescents

SUMMARY:
"Hoarding "is a common behavior among Holocaust survivors and is related to the traumatic events they have experienced, and we assume that storage behavior and eating disorders are related to future generations of Holocaust survivors.

ELIGIBILITY:
Inclusion Criteria:

1. Jewish Holocaust survivors living in Germany and Israel who have expressed their written and written consent to participate in monitoring and testing, and who are able to answer the research questionnaires.

   • Their direct offspring and their children (second and third generation)
2. The control population - non-Jewish subjects who are not the descendants of Holocaust survivors living in Germany who have expressed their written and oral consent to participate in monitoring and testing and who are able to answer the research questionnaires and whose parents were not imprisoned in the camps second.

Exclusion Criteria:

* (Participants who do not agree to participate (did not sign informed consent form
* Respondents who are unable to answer interviewer questions
* Non-Jewish subjects whose parents were in camps (ie prisoner camps, labor camps, etc.) during the second war.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Jewish Holocaust survivors living in Germany and Israel Their direct offspring and their children (second and third generation)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Hoarding | Three years
  Questionnaire that will follow behaviour over generations